CLINICAL TRIAL: NCT02392923
Title: Quality of Life and Body Functions in a Representative Swedish Population
Brief Title: Quality of Life in a Representative Swedish Population
Acronym: Normalen
Status: Completed | Type: Observational
Sponsor: Eva Haglind (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Eva Haglind, Professor, Consultant Surgeon, Göteborg University
Organization: Göteborg University (Other)
Other Study IDs: QoL normal Swedes
Record Dates: First submitted 2014-06-18; First posted 2015-03-19 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Quality of Life
Keywords: health related quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cohort descriptive study of quality of life and body functions in a reference population of Swedish inhabitants from age 30 to age 89. The population was selected to be representative for the general Swedish population and 500 in each 10 year group, 250 men and 250 women.

The population is contacted and asked for informed consent, whereafter a questionnaire of about 200 questions, used in a number of studies in clinical studies and trials, are sent out.

The results will be used as reference values to our patient cohorts

DETAILED DESCRIPTION:
Individuals contacted by letter with information about the study and it's aim. The next step is a telephone contact from the study secretariate where the person can ask for more detailed information and put questions to the reserach nurse. The call leads up to a question to the person, if the questionnaire can be sent. If yes, the questionnaire is posted includeing the consent form and an pre-paid return envelope. After two weeks a thank you/reminder letter is sent out, and if no reply one more phone call is made two weeks further on.

ELIGIBILITY:
Inclusion Criteria:

* list generated by the equivalent to inland revenue ("Skatteverket", Sweden)

Exclusion Criteria:

* unable to read and understand Swedish
* no informed consent

Ages: 30 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Swedish cohort aged 30-89, representatvie for entire Swedish population age 30 -89
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
quality of life | 12 months
  answers to specific questions in questionnaire The time frame of most questions is "How would you rate your quality fo life during the last month"

SECONDARY OUTCOMES:
sexual health | 12 months
  answers to various questions in questionnaire
gastrointestinal function | 12 months
  answers to various questions in questionnaire
urinary function | 12 months
  answers to various questions in questionnaire
other body functions | 12 months
  answers to various questions in questionnaire
mental health | 12 months
  answers to various questions in questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eva Haglind, Principal Investigator — Department of Surgery, Institure for Clinical Sciences, Sahlgernska Academy at Göteborg University
Locations (1):
- Göteborg University, Sahlgrenska Academy, Inst Clinical Sciences, Dept Surgery,, Gothenburg, Sweden

REFERENCES:
- [Derived] Bock D, Angenete E, Gonzales E, Heath J, Haglind E. Assessing health, quality of life and urogenital function in a sample of the Swedish general population: a cross-sectional study. BMJ Open. 2018 May 5;8(5):e021974. doi: 10.1136/bmjopen-2018-021974. PMID 29730632